CLINICAL TRIAL: NCT02112539
Title: Pivotal Study of the AggreGuide A-100 Adenosine Diphosphate (ADP) Assay to Evaluate the Effect of ADP Blocking Drugs on Platelet Aggregation on the AggreGuide A-100 Instrument
Brief Title: Aggreguide A-100 ADP Assay Evaluation
Status: Completed | Type: Observational
Sponsor: Aggredyne, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Val 0072-B
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Platelet Aggregation; ADP Blockers
MeSH Terms: interventions — Platelet Aggregation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADP Blockers: platelet aggregation in response to antiplatelet drugs
  Interventions: Other: platelet aggregation measurement

INTERVENTIONS:
Other: platelet aggregation measurement

SUMMARY:
The study is to characterize the AggreGuide ADP Assay's performance.

ELIGIBILITY:
Inclusion Criteria:

* 18-75

Exclusion Criteria:

* less than 60 kg
* on antiplatelet meds other than aspirin
* antiplatelet drugs contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Platelet Activity Index (PAI) | 1 week
  PAI at baseline and after taking ADP blocking antiplatelet drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Teitel, MD, Principal Investigator — Unafilliated
Locations (1):
- Juno Research, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No